CLINICAL TRIAL: NCT03373084
Title: Imaging Location of Hamstring Muscle Lesions in Sport and Relationships With Injury Mechanism.
Acronym: HAMMER
Status: Terminated | Type: Observational
Why Stopped: Reduced recruitment potential for study participants.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1708231; ANSM (Other: 2017-A03433-50)
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Sport Injury; Hamstring Muscle Lesions
Keywords: Magnetic Resonance Imaging (MRI); Ultrasound; Sport; Hamstring muscle; Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hamstring muscle lesions: Patients with hamstring muscle lesions in sport will be included. As usual practice they will have Magnetic Resonance Imaging (MRI) or ultrasound, and will answer to self-questionnaire
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: ultrasound; Other: Self-questionnaire

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) or ultrasound will be performed to determinate location of the lesion
Other: ultrasound — Magnetic Resonance Imaging (MRI) or ultrasound will be performed to determinate location of the lesion
Other: Self-questionnaire — Self-questionnaire will be completed by patient. In this questionnaire patients will describe the circumstances of the injury and their personal characteristics and level of sporting practice.

SUMMARY:
Hamstring muscle injuries are a common pathology in sports mainly present in sprint and acceleration sports, accounting for about 12% of all football injuries. Because of their frequency, risk of reinjury and financial cost, they can be considered as a public health problem. Improving knowledge of the pathophysiology of hamstring muscle injury appears to be a relevant research focus for prevention purposes.

DETAILED DESCRIPTION:
This study is a cohort of athletes in the context of suspicion of hamstring muscle injuries.

ELIGIBILITY:
Inclusion Criteria:

* To be recreational sportsmen, competitions, amateurs, high-level or professional
* Aged 18 to 50 years
* Perform an Magnetic Resonance Imaging (MRI) or an ultrasound of the thigh in the context of the suspicion of an acute hamstring muscle injury
* Injury during sport since less 21 days old.

Exclusion Criteria:

* a history of surgery of the anterior cruciate ligament with removal of the transplant in the posterior compartment of the thigh
* an antecedent of surgery of the thigh.
* inability to understand the French language for completing the self-questionnaire

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Athletics with thigh injury will be included.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
location of the lesion of injury | at inclusion
  Correlation between location of the lesion and mechanism of onset of injury. Location of the lesion will be measured by Magnetic Resonance Imaging (MRI) or ultrasound results. For location of the lesion, it is a combination of the injured muscle, damaged tissue and the area in the posterior compartment of the thigh.
mechanism of onset of injury | at inclusion
  Correlation between location of the lesion and mechanism of onset of injury. Location of the lesion will be measured by Magnetic Resonance Imaging (MRI) or ultrasound results.
  Mechanism of onset of injury will be check by self-questionnaire.

SECONDARY OUTCOMES:
mapping of hamstring lesions | at inclusion
  Analyzed of mapping of hamstring lesions with Magnetic Resonance Imaging (MRI) / ultrasound.
  Compare the MRI and ultrasound maps and the performance of the two means to determine the location of the lesion.
volumetric analysis of the hamstrings | at inclusion
  A standardization of the images to allow a better comparison between individuals

CONTACTS AND LOCATIONS:
Overall Officials: Pascal EDOUARD, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No